CLINICAL TRIAL: NCT01994928
Title: Prospective Randomised Study on Preoxygenation in the Intensive Care Unit Using a Nose-mouth Mask Versus High Flow Nasal Cannula Oxygen.
Brief Title: Preoxygenation in the Intensive Care Unit Using a Nose-mouth Mask Versus High-flow Nasal Cannula Oxygen.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Stefan Kluge, Prof. Dr. Stefan Kluge, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PV-4429
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Intubation

ARMS (2):
- Nose-mouth mask (Active Comparator): Performance of intubation after preoxygenation using a nose-mouth mask.
  Interventions: Device: Nose-mouth mask; Procedure: Intubation
- High flow nasal cannula oxygen (Experimental): Performance of intubation after preoxygenation using high flow nasal cannula oxygen.
  Interventions: Device: High flow nasal cannula oxygen; Procedure: Intubation

INTERVENTIONS:
Device: Nose-mouth mask — Preoxygenation using a nose-mouth mask.
  Arms: Nose-mouth mask
Device: High flow nasal cannula oxygen — Preoxygenation using high flow nasal cannula oxygen.
  Arms: High flow nasal cannula oxygen
Procedure: Intubation — Intubation

SUMMARY:
Preoxygenation is routinely performed before endotracheal intubation. In the intensive care unit, preoxygenation is often accomplished using a nose-mouth mask. It seems probable that high flow nasal cannula oxygen, which is used in the treatment of patients with hypoxemic respiratory failure, is equally effective in preventing the development of hypoxemia during intubation. In this prospective randomized study preoxygenation using high flow nasal cannula oxygen is compared with preoxygenation via nose-mouth mask in patients with hypoxemic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* patients treated in an intensive care unit
* indication for intubation
* presence of hypoxemic (SaO2/fraction of inspired oxygen(FiO2): 300 or less) respiratory failure
* informed consent

Exclusion Criteria:

* blocked nasopharynx
* contraindications for nose-mouth mask or high flow nasal cannula oxygen
* expected difficult airway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Mean decrease in the saturation of oxygen (SpO2) during intubation. | during intubation
  Mean decrease in the saturation of oxygen measured by pulse oximetry (SpO2 [%]) during intubation.

SECONDARY OUTCOMES:
Changes in blood gases after intubation. | 30 minutes after intubation
  Changes in arterial blood gases collected from arterial line (PaO2/FiO2 [mmHg] and PaCO2 [mmHg]) after intubation.

OTHER OUTCOMES:
Changes in hemodynamics. | during intubation and up to 30 minutes after intubation
  Changes in mean arterial pressure [mmHg] measured via arterial line.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Department of Intensive Care Medicine, Hamburg, Germany

REFERENCES:
- [Result] Simon M, Wachs C, Braune S, de Heer G, Frings D, Kluge S. High-Flow Nasal Cannula Versus Bag-Valve-Mask for Preoxygenation Before Intubation in Subjects With Hypoxemic Respiratory Failure. Respir Care. 2016 Sep;61(9):1160-7. doi: 10.4187/respcare.04413. Epub 2016 Jun 7. PMID 27274092